CLINICAL TRIAL: NCT04786886
Title: Patient Performance and Acceptance of Virtual Reality Visual Field Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Alana L Grajewski, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20190679
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Visual Field Defect, Peripheral; Visual Field Defect, Nasal Step; Visual Field Defect, Paracentral Scotoma of Both Eyes
Keywords: Retinal Sensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual Reality Visual Field Group (Experimental): Participants in this group will have virtual reality visual field testing during standard of care follow-up visit.
  Interventions: Other: VIrtual Reality Visual Field Exam

INTERVENTIONS:
Other: VIrtual Reality Visual Field Exam — Virtual reality visual field exam will be administered using the virtual reality headset. Exams can take up to 20 minutes.

SUMMARY:
The purpose of this research is to study the effectiveness and patient experience when measuring visual fields using virtual reality goggles.

ELIGIBILITY:
Inclusion Criteria:

* Any patient >13 years old at Bascom Palmer Eye Institute
* Patients who either have glaucoma, are glaucoma suspects, or have a strong family history of glaucoma

Exclusion Criteria:

* Adults unable to consent, pregnant women, prisoners
* Patients under the age of 13

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Operational Effectiveness | Day 1
  Operational effectiveness will be reported as the length of the visit and virtual reality visual field exam testing times. Both will be measured in minutes.
Medical Effectiveness as Measured by Visual Field Indexes | Day 1
  Medical effectiveness will be evaluated by visual field indexes, such as mean deviation, pattern standard deviation, and foveal threshold, which are all measured in decibels. These values are generated based on the participants' performance in the visual field exam.
Medical Effectiveness as Measured by Glaucoma Hemifield Test | Day 1
  Medical effectiveness will be evaluated by the glaucoma hemifield test. This value is generated based on the participants' performance in the visual field exam.
Reliability Indices | Day 1
  Reliability index is generated based on the participants' performance in the visual field exam.

CONTACTS AND LOCATIONS:
Overall Officials: Alana Grajewski, MD, Principal Investigator — University of Miami
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No